CLINICAL TRIAL: NCT04382495
Title: Impact of COVID-19 Pandemic on Cancer Care Provision: a Cross-sectional Study of Egyptian Patients' Perspectives and Concerns
Brief Title: The Impact of COVID-19 Pandemic on Cancer Care
Status: Completed | Type: Observational
Sponsor: El Zaitoun Specialized Hospital (Other Government)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Aalaa Abdou, Principle Investigator, El Zaitoun Specialized Hospital
Other Study IDs: Cancer Care during Covid-19
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cancer
Keywords: Cancer Care; COVID-19
MeSH Terms: conditions — Neoplasms; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — online survey

SUMMARY:
The situation of COVID-19 pandemic creates many challenges for cancer patients and caregivers. Some modifications in cancer management have been evolved from cancer societies and organizations to support oncology professionals as much as possible to deliver optimal care to their cancer patients in such exceptional circumstances, and to protect patients from infection with COVID-19 as much as possible.

DETAILED DESCRIPTION:
In oncology practice during this pandemic, many cancer patients still feeling uncertainty about their cancer management and treatment outcome . The study is aiming to better understand the impact of the COVID-19 pandemic on cancer care from patients' and survivors' perspective.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients or survivors in Egypt.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study survey will be distributed through social media to cancer patients and survivors in Egypt. We plan to enroll as many participants as possible without limitation of the number although we hope to achieve at least 400 participants.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
patients' and survivors' perspective of their cancer care during COVID-19 pandemic | one month
  measured by online survey to understand the impact of COVID-19 pandemic on cancer care

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelaziz, MD, Study Director — Ain Shams University
Locations (1):
- EgyBrit Medical Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
email